CLINICAL TRIAL: NCT03381053
Title: Prospective Multicenter Cohort Study to Compare Pathologic Type, NIH and WHO Criteria, and Mechanism of GIST Malignant Transformation
Brief Title: Study to Compare Pathologic Type, NIH and WHO Criteria,and Mechanism of GIST Malignant Transformation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Ruijin Hospital (Other); Fudan University (Other); Changhai Hospital (Other); Shanghai Changzheng Hospital (Other); Huashan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SH-GIST2017pathology
Record Dates: First submitted 2017-12-18; First posted 2017-12-21 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Method of Differentiating Benignancy and Malignancy, Grading and Staging for GIST
Keywords: GIST; Grading and Staging
MeSH Terms: conditions — Neoplasms | interventions — Imatinib Mesylate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment observation group: According to the morphological criteria, the NIH scheme, and the WHO standard, GIST patients are divided into two groups, benign group and malignant group. In fully informed of their illness, patients are free to choose the sequence treatments according to their own gene mutation status and economic conditions. Patients who choose postoperative Imatinib treatment are labeled treatment group.
  Interventions: Drug: Imatinib 400mg
- Control observation group: According to the morphological criteria, the NIH scheme, and the WHO standard, GIST patients are divided into two groups, benign group and malignant group. In fully informed of their illness, patients are free to choose the sequence treatments according to their own gene mutation status and economic conditions. Patients who choose no Imatinib treatment are labeled observation group.

INTERVENTIONS:
Drug: Imatinib 400mg — The NIH assessment of patients with surgical excision of GIST with moderate to high risk of recurrence was recommended imatinib 400mg treatment.
  Groups: Treatment observation group

SUMMARY:
Evaluate the reliability of morphology standards for GIST pathologic type, staging and grading by retrospective analyzing clinical data; on this basis, establish a GIST standardized and individualized treatment mode to maximum benefit GIST patients, avoid under- and over-treatment

DETAILED DESCRIPTION:
1. Retrospective analysis of GIST cases in the recent five years: the GIST clinical data of Fudan University Zhongshan Hospital from 2007 January to 2012 December were collected. By reviewing the HE slides, GIST was evaluated by 12 indicators, NIH scheme and WHO standard. Accomplish the gene sequencing of KIT, PDGFRA, B-raf, and SDH. Follow up the patients about their treatment and prognosis. Analyze and compare the advantages and disadvantages of the histomorphology indicators, NIH scheme, and WHO standard.
2. Organize the first multicenter prospective cohort study of GIST individualized treatment based on the histomorphology. Obtain the evidence of histological assessment for GIST by following up patients for 3 years.
3. Establish an evaluation criteria based on the morphology of GIST. Make objective evaluations about GIST tumor size, tumor location and gene mutation status in the prognosis estimate. Make rules to effectively guide individualized treatment of GIST.

ELIGIBILITY:
Inclusion Criteria:

* All patients pathologically diagnosed with GIST during the period from 2017 to 2020

Exclusion Criteria:

* Only have Biopsy diagnosis
* Only have Liver metastasis or peritoneal dissemination
* Received imatinib treatment before surgery

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with GIST by pathology
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with tumor recurrence | 3 years
Number of participants with tumor metastasis | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Hou Ying Yong, Doctor, Study Chair — Shanghai Zhongshan Hospital
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No